CLINICAL TRIAL: NCT04678219
Title: A Pilot Study Examining a Vegan/Low-Sulfur Diet Versus the Specific Carbohydrate Diet in Patients With Primary Sclerosing Cholangitis
Brief Title: A Pilot Study Examining Diet in Primary Sclerosing Cholangitis
Acronym: DINER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of California, Davis (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Joshua Korzenik, Director, Crohn's and Colitis Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002075
Record Dates: First submitted 2020-08-18; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: Primary Sclerosing Cholangitis; Diet; Specific Carbohydrate Diet; Low-Protein; Low-Sulfur; Vegan
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: 20 subjects will be randomized onto either the Specific Carbohydrate Diet or the low-protein (vegan/low-sulfur) diet, with 10 subjects per diet.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-Protein/Vegan/Low-Sulfur Diet (Experimental): This is a specific diet that is both vegan and low in protein. The vegan diet eliminates all animal products, (including meats, eggs, dairy products) and animal by-products such as honey.
  Interventions: Other: Dietary Intervention
- Specific Carbohydrate Diet (Experimental): The Specific Carbohydrate Diet emphasizes consumption of specific carbohydrates that require minimal digestion. Therefore, it eliminates most carbohydrates, including grains, starches, dairy and sugars.
  The idea behind this diet is that it reshapes the microbiome of the intestines. The diet restricts the intake of certain carbohydrates that may increase the growth of "bad" bacteria possibly contributing to inflammation. By restricting the amount of these carbohydrates in the microbiome, the diet aims to reduce their activity in the gut and reduce inflammation.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Subjects will be placed on 1 of 2 diets for a treatment period of 8 weeks with the support of dietitians; it will then be evaluated whether they can continue this diet on their own for 4 weeks.

SUMMARY:
This research study is exploring the effects of dietary intervention in PSC. Study participants will be randomly assigned to either the Specific Carbohydrate Diet (SCD) or a vegan/low-sulfur diet for 8 weeks; the entire study will last approximately 14 weeks. Participants will work with BWH Registered Dieticians and receive dietary educational materials, recipes, and a food procurement stipend to support the new diet. Subjects will attend 7 video visits and have regular lab tests performed, requiring blood and stool samples.

DETAILED DESCRIPTION:
The chronic, autoimmune liver disease Primary Sclerosing Cholangitis (PSC) is a progressive cholestatic, hepatobiliary disease characterized by inflammation and fibrosis of the bile duct. As the disease progresses, it may result in debilitating bile duct cirrhosis, malignancy, and liver failure. Although the list of drugs studied for the treatment of PSC is extensive, the main, and commonly only, treatment option remains liver transplantation. Dietary manipulation is an approach of high interest to patients. Presumably, diet may have some influence on the intestinal microbiome and have a modifying impact on the diseases but this has not been well established.

The investigators propose a study period of approximately 14 weeks to evaluate the effects of the SCD and vegan/low-sulfur diet on the intestinal microbiome and bile acid composition in stool and serum. Patients will visit their study site or participate in a video visit 7 times over the course of the study. At the screening visit (Week 0), eligibility will be assessed, lab tests will be performed, and subjects will be randomized to dietary instruction on one of the two diets with educational materials, recipes, and food procurement stipend provided. Consent will be signed at or before the screening visit either in-person or remotely. Patients will be asked to collect a stool sample and complete a Food Frequency Questionnaire (FFQ).

The treatment phase of 8 weeks will begin at the baseline visit (Week 2). At each of the four time points during the treatment phase (Week 4, 6, 8, 10), participants will record in real-time what they eat by a smartphone app for 3-days, one of which includes a weekend. To enhance compliance to the intervention protocol, the dedicated study coordinator along with the Registered Dietitian will review the food diary data in real-time and discuss any challenges to comply with the meal intervention. After the 8-week treatment period is complete, patients will be encouraged to continue with their diet, self-directed, for 4 weeks following the end of the treatment phase (Week 10). Subjects will be asked to return for one final visit at Week 14 to complete a 3-day food diary and have labs drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between 18 and 70 years of age, inclusive based on the date of the screening visit
2. Willing and able to give informed consent prior to any study specific procedures being performed
3. Diagnosis of PSC documented by typical cholangiogram findings with no evidence of a secondary cause of sclerosing cholangitis
4. Serum alkaline phosphatase greater than 1.5 times the upper limit of the normal (ULN) reference range
5. Simple clinical colitis activity index < 5
6. For subjects on UDCA, the dose of UDCA must have been stable for at least 3 months before screening. For subjects not on UDCA, no UDCA use for at least 3 months before screening.
7. Platelet count > 150,000/mm3
8. Albumin > 3.3 g/dL
9. Serum creatinine < ULN
10. Willing and able to comply with scheduled visits, laboratory tests, stool collection, and other study procedures including to follow a vegan/low-sulfur diet or SCD for the duration of the trial regardless of treatment arm randomization
11. Able to read English and complete PSC PRO independently

Exclusion Criteria:

1. Pregnant or lactating females
2. ALT > 10 x ULN
3. Total bilirubin > 2 X ULN
4. INR > 1.2
5. Decompensated cirrhosis defined by ascites, hepatic encephalopathy, or variceal bleeding
6. Small duct PSC
7. Other causes of liver disease including secondary sclerosing cholangitis, viral, metabolic, alcoholic, and other autoimmune liver diseases. Subjects with non-alcoholic fatty liver disease may be included if there is no evidence of NASH in the opinion of the investigator
8. Positive AMA
9. History of liver transplantation
10. History of hepatocellular carcinoma or cholangiocarcinoma
11. Ascending cholangitis within 90 days of enrollment
12. Any antibiotic use within 90 days of enrollment or planned antibiotic use during the study period
13. Current vegetarian or adherence to the SCD
14. Nut allergy (Many of the recipes included in the specific carbohydrate diet substitute nut flour for wheat flour. Subjects randomized to either the specific carbohydrate diet arm will have difficulty with dietary adherence as they will be intolerant of this dietary staple).
15. Inability to complete dietary log.
16. History of malignancy within 5 years except for adequately treated carcinoma in situ of the cervix and basal or squamous cell carcinoma.
17. Concurrent participation in another therapeutic clinical trial
18. Celiac disease
19. Any laboratory abnormality or condition which in the opinion of the investigator could adversely affect the safety of the participant or impair the assessment of the study results

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Shannon index | Control period (Weeks 0-2) to Week 14
  The primary endpoint will be the within group change in the Shannon diversity index. The Shannon diversity index is used to characterize species diversity in a community (the diversity in the fecal microbiome).

SECONDARY OUTCOMES:
ALP level | Control period (Weeks 0-2) to Week 14
  The investigators will be evaluating the trend of alkaline phosphatase reduction (U/L).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Korzenik, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States